CLINICAL TRIAL: NCT03438526
Title: Better Outcome With Melatonin Compared to Placebo Administered to Normalize Sleep-wake Cycle and Treat Hypoactive ICU Delirium The Basel BOMP-AID Randomized Trial
Brief Title: The Basel BOMP-AID Randomized Trial
Acronym: BOMP-AID
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKNZ 2018-00161
Record Dates: First submitted 2018-01-29; First posted 2018-02-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hypoactive Delirium
MeSH Terms: interventions — Melatonin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Circadin ®) (Experimental)
  Interventions: Drug: Melatonin (Circadin ®)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin (Circadin ®) — 4 mg of oral melatonin at 8 p.m. for the length of the duration of the hypoactive delirium
  Arms: Melatonin (Circadin ®)
Drug: Placebo — Lactose monohydrate, cellulose powder, magnesium stearate (Ph. Eur.), mocrocristalline cellulose
  Other Names: Oral tablet
  Arms: Placebo

SUMMARY:
Delirium is a neurobehavioural syndrome that frequently develops in the postoperative and/or ICU setting. The incidence of elderly patients who develop delirium during hospital stay ranges from 11-82%. Delirium was first described more than half a century ago in the cardiac surgery population, where it was already discovered as a state that might be accompanied by serious complications such as prolonged ICU and hospital stay, reduced quality of life and increased mortality. Furthermore, the duration of delirium is associated with worse long-term cognitive function in the general ICU population. This long-term experience with delirium suggests a high socioeconomic liability and has been a focus of many studies. The aforementioned consequences of delirium are observed in all of three subtypes: hypoactive, hyperactive, and mixed. Pharmacological treatment options for hypoactive delirium are lacking. Since patients in hypoactive delirium suffer from disturbed circadian rhythm, the investigators suggest that the administration of melatonin as a promising possibility in these patients to shorten delirium duration and to lower its severity. Previous investigations confirmed loss of melatonin rhythm in patients that had developed delirium thus reasoning the study hypothesis.

In this randomized study, the investigators aim to test the hypothesis that the reinstitution of a normal circadian rhythm by the administration of melatonin compared to placebo after diagnosis of hypoactive delirium, decreases the duration of delirium and reduces the transmission to a form of agitated delirium. The administration might have to be repeated several times to achieve resolution of delirium.

DETAILED DESCRIPTION:
Delirium is a neurobehavioural syndrome that frequently develops in the postoperative and/or ICU setting. The incidence of elderly patients who develop delirium during hospital stay ranges from 10-80%. Delirium was first described more than half a century ago in the cardiac surgery population, where it was already discovered as a state that might be accompanied by serious complications such as prolonged ICU and hospital stay, reduced quality of life and increased mortality. Furthermore, the duration of delirium is associated with worse long-term cognitive function in the general ICU population. This long-term experience with delirium suggests a high socioeconomic liability and has been a focus of many studies. Due to the multifactorial origin of delirium, there are several but no incontestable options for prevention and symptomatic treatment. Overall, delirium represents a high burden not only for the patient and his/her family members, but also for the medical care team that aims to prevent postoperative delirium to avoid serious consequences associated with it.

The aforementioned consequences of delirium are observed in all of three subtypes: hypoactive, hyperactive, and mixed. Many studies have been conducted to prevent and treat hyperactive and mixed delirium. Hypoactive delirium, suggested to be the most frequent form of delirium, is a different case: as it corresponds to a patient that is calm and as such doesn't cause any harm or inconvenience to himself or the caring medical team it also leads to two major problems. First, it is already known that hypoactive delirium is hard to detect. Second, because hypoactive delirious patients are calm or even asleep most of the time this delirium subtype doesn't go along with the same urge to become active in order to prevent harm. Also, pharmacological treatment usually addresses hyperactive and mixed delirium in standard operating procedures, whereas treatment of hypoactive delirium remains supportive. Pharmacological treatment options for hypoactive delirium are lacking. Since patients in hypoactive delirium suffer from disturbed circadian rhythm, investigators suggest that the administration of melatonin is a promising possibility in these patients to shorten delirium duration and to lower its severity. Previous investigations confirmed loss of melatonin rhythm in patients that had developed delirium thus reasoning the study hypothesis. Of note, melatonin is to be investigated for ICU delirium prevention in an Australian study, as the potential of chronotherapy to reduce delirium incidence has been suggested in a recently published article. The administration of dexmedetomidine to treat the disturbed circadian rhythm in hyperactive and mixed delirious ICU patients will be investigated in one of the investigators' current studies, but because of its sedative nature it clearly doesn't represent a treatment option for hypoactive delirium.

The aim of the BOMP-AID trial is to assess the superiority of melatonin to placebo for the treatment of hypoactive delirium in the ICU. The study hypothesis is based on the assumption that melatonin compared to placebo (Lactose monohydrate, cellulose powder, magnesium stearate (Ph. Eur.), mocrocristalline cellulose) administered at night restores a normal circadian rhythm, thus decreasing the duration of delirium and reducing the transmission to a form of agitated delirium.

Investigators would like to recruit 190 patients right after the diagnosis of hypoactive delirium. The administration might have to be repeated several times to achieve resolution of delirium.

After the first administration of melatonin or placebo at 8 p.m. investigators shall follow the standard operating procedure for hypoactive delirium for further treatment of delirium during daytime. In case of previously undiagnosed mixed delirium investigators are forced to follow the standard operating procedure for mixed delirium that includes the administration of haloperidol, quetiapine or trazodone. During the consecutive nightly hours the randomized study substance will be administered again if indicated. The latter will allow investigators to clearly detect the suggested shortening of delirium duration in the cohort where melatonin is being used as treating agent. Any use of drugs to treat forms other than hypoactive will be recorded.

The primary outcome measure is delirium duration in shifts of 8 hours each. Due to difficult diagnosis of hypoactive delirium, the investigators will consider those with an ICDSC score > 2 (subsyndromal delirium) and Richmond Agitation Sedation Scale (RASS) score < 0 in absence of induced coma as eligible for study inclusion. If patients reveal an ICDSC score > 2 and a RASS score < 0 a member of the study team will assess the patient according to DSM-V delirium criteria REF] for definite study inclusion. The end of the delirium will be deﬁned as the end of the last shift with an ICDSC > 2 and a RASS score < 0 that precedes a minimum of two subsequent shifts with an ICDSC < 3.

Secondary outcomes can be listed as follows:

* Delirium-free days at 28 days after study inclusion
* Death until day 28, day 90, and day 365 from ICU admission
* Number of ventilator days
* Length of ICU stay (hours)
* Length of hospital stay (days)
* Sleep quality, assessed by the Richards-Campbell Sleep Questionnaire (RCSQ; total score)

Since melatonin has no known major side effects evidence of its way of function in the human body strongly suggests high benefit for treatment of hypoactive delirium going along with increased comfort and safety also for critically ill patients. No severe adverse events are expected by its use in delirious patients after careful enrolment following investigators exclusion criteria.

Other outcome measures:

The following outcomes are measured by smartwatches. The smartwatches will be attached half an hour before the administration of the drug (07:30 p.m.) and left attached as long as possible, but at least until 6 a.m. of every day of the study period.

The following smartwatch assessments are based on activity (counts/min):

* Sleep duration per night (minutes) defined as the period from lights off to lights on
* Number of sleep interruptions (number of consecutive 5-min bouts of >0 activity)
* The relative amplitude (RA) calculated from the ratio of the most active 10-hour period (M10) to the least active 5-hour period (L5) across the averaged 24-hour profile (assessment depends upon patient cooperation during the day with keeping the smartwatch attached)
* Interdaily stability (IS), which quantifies the invariability day by day, that is, how well the sleep-wake cycle is synchronized to supposedly stable environmental cues. Timing information comes from determining the onset of the 5 hours with least activity (L5 onset) and onset of the 10 hours with most activity (M10 onset).

In addition, wrist/skin temperature (degrees/min) will be registered to assess degree of relaxation (i.e., difference in degrees Celsius per minute between distal skin regions (finger, feet etc) and proximal skin regions (clavicular, sternum etc).

Follow-up:

To assess long-term follow-up of patients who received melatonin and compare it to those who received placebo, we will perform a follow-up at three and twelve months after the prevailing hospital case has been officially closed (discharge date). With this follow-up, we will assess the following information equally at three and twelve months (information either given by the patient or his/her family/contact person):

* Death after hospital discharge
* Hospital readmission
* Activities of Daily Living Questionnaire (ADLQ)
* Additional episodes of delirium after study closeout

CRF assessments:

On our electronic case report form, we will document the following information concerning our study participants (sequential order):

* Patient information including socioeconomic status
* Study group
* Study eligibility
* Results of the planned assessment tools
* Cardiovascular parameters
* Lab values
* Drugs administered
* Nursing interventions
* Outcome overview
* Follow-up at three and twelve months

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Adult patients (aged 55 years or older)
* Current delirium (hypoactive type) detected by a specialised assessment method: ICDSC score >2 and RASS score < 0

Exclusion Criteria:

Participants meeting the following criteria are excluded from the study:

* Delirium prior to ICU admission
* Sleep disorder not caused by hypoactive delirium
* Sedation in the ICU
* Hypersensitivity to the studied substances (i.e., melatonin, placebo content)
* Age <55 years
* Terminal state
* Status epilepticus or postictal states following seizures on electroencephalogram (EEG)
* Active psychosis
* Substance abuse in current medical history
* Dementia
* Pregnancy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Duration of hypoactive delirium | From study inclusion to delirium resolution, assessed daily until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 28 days
  Duration of hypoactive delirium in the ICU in 8-hour shifts

SECONDARY OUTCOMES:
Delirium-free days at 28 days after study inclusion | From study inclusion to ICU discharge, assessed up to 28 days
  Duration of Delirium-free days measured in days
Death until day 28, day 90, and day 365 from ICU admission | Assessed at 28 days, 90 days, and 365 days after study inclusion
  Telephone Survey 28 days, 90 days and 365 days after study inclusion
Number of ventilator days | From study inclusion until ICU discharge, assessed daily until the date of withdrawal of mechanical ventilation or date of death from any cause, whichever came first, assessed up to 28 days
  Number of days on mechanical ventilation measured in days
Length of ICU stay | From ICU admission to ICU discharge, assessed daily until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 28 days
  Length of ICU stay measured in hours
Length of hospital stay | From hospital admission to hospital discharge, assessed daily until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 90 days
  Length of hospital stay measured in days
Sleep quality | From study inclusion until study termination, assessed daily until the date of first documented progression (i.e., delirium resolution) or date of death from any cause, whichever came first, assessed up to 28 days
  Assessed by the Richards-Campbell Sleep Questionnaire (RCSQ; total score)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Hollinger, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Study results will be communicated to patients based on expected speed-up in convalescence from delirious state. During the study ongoing and until publication there will be no access to our data.

REFERENCES:
- [Derived] Hollinger A, von Felten S, Sutter R, Huber J, Tran F, Reinhold S, Abdelhamid S, Todorov A, Gebhard CE, Cajochen C, Steiner LA, Siegemund M. Study protocol for a prospective randomised double-blind placebo-controlled clinical trial investigating a Better Outcome with Melatonin compared to Placebo Administered to normalize sleep-wake cycle and treat hypoactive ICU Delirium: the Basel BOMP-AID study. BMJ Open. 2020 Apr 30;10(4):e034873. doi: 10.1136/bmjopen-2019-034873. PMID 32354780